CLINICAL TRIAL: NCT00088361
Title: The Effects of Respiratory Motion on CT Based Attenuation Correction of Positron Emission Tomography Data: Liver and Heart Studies
Brief Title: Effect of Respiratory Motion on Positron Emission Tomography Imaging
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040237; 04-CC-0237
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-06

CONDITIONS: Healthy; Tomography; Emission Computed
Keywords: Reconstruction; PET Artifacts; PET/CT Motion Artifacts; Liver; Heart; Respiratory Motion

SUMMARY:
This study will determine how breathing motions may affect positron emission tomography (PET) scans. It has been discovered that the quality of PET scans varies according to which part of the breathing cycle patients hold their breath.

NIH Clinical Center patients 12 years of age and older who are scheduled to have PET and computed tomography (CT) scans as part of their standard medical care may be eligible for this study.

Participants have their scheduled PET or CT scan as they normally would and are asked to hold their breath after breathing out, as is usual. In addition, for this study, patients are also asked hold their breath after breathing in and again at a point between breathing in and out. Each breath-hold is for around 15 seconds. The scans for each of the three different breath-holds are examined for differences.

Some patients may also be asked to breathe through a tube called a pneumotachometer, or spirometer, to determine their normal breathing pattern. This involves breathing through a mouthpiece similar to a snorkel mouthpiece and takes about 2 minutes.

DETAILED DESCRIPTION:
Current clinical FDG imaging with the NIH's PET/CT machine (and in fact with most commercial PET/CT machines) requires a CT scan be acquired prior to the PET scan. This CT scan is used for attenuation correction of the PET data and to permit fusion of anatomical and metabolic image data.

One difficulty with use of the CT scan for attenuation correction ('CTAC') is that the CT scan is rapid compared to the breathing cycle. Each CT slice captures the lungs at one (usually arbitrary) phase of the respiratory cycle. The PET data on the other hand take many minutes to acquire, and so average the motion effects of the entire respiratory cycle together. This 'freezing' of the respiratory cycle by the CT, and blurring of the respiratory cycle during PET produces a mis-match between the PET and CT data. This mis-match can produce improper attenuation correction during PET reconstruction, especially at soft tissue/lung interfaces. The existence of this phenomenon has been reported in the literature [1-7], especially at the dome of the liver, but it has not been thoroughly quantified. Little or no data is available to indicate the quantitative errors the effect produces in cardiac imaging[8]. This despite the fact that the myocardium is only about 10mm thick, and it has been reported that the heart moves on average 9mm (and as much as 14mm) during a single average respiratory cycle[9].

The purpose of this protocol is to determine the degree to which respiratory motion may influence quantitative PET imaging, especially at the lung/liver interface and free wall of myocardium. By characterizing the magnitude of the effect, we hope to gain knowledge about when correction for the effect is and is not necessary. It is hoped that the information gained will also allow us to suggest potential methods to perform such corrections.

To gain the above information we will modify the CT acquisition protocol for subjects already scheduled to undergo a whole body FDG PET/CT scan. In summary, rather than acquiring the usual single full radiation exposure CT (taking approx 20-30 seconds), we will acquire 3 CT scans (each taking approximately 20-30 seconds), each at 1/3 the usual radiation exposure. Each CT will be acquired at a different phase of the respiratory cycle (as opposed to current acquisition, which is only at end-expiration). The subsequent PET data will be acquired as usual, but will be processed and analyzed separately with each of the CT scans and also with a summed CT scan.

Note that subjects agreeing to participate in this protocol will receive no additional radiation exposure. Participation in the protocol will extend the current overall scan time (typically greater than 45 minutes) a very small amount (about 40-60 additional seconds for imaging, and about 60 additional seconds for patient set up, etc).

ELIGIBILITY:
* INCLUSION CRITERIA

Up to 30 subjects will take part in the study, chosen from sequential incoming clinical patients who are scheduled for PET/CT studies of the torso and who have had or will have a diagnostic CT within one week of the PET/CT study, without regard to disease. The number of subjects selected for study per week will depend on patient load and availability of scanner and technologist). Approximately an equal number of males and females will be selected by alternating each selection between male and female. The selection of subjects asked to participate will be random, in the sense that whenever technologist and analysis time is available, the next subject scheduled for a whole body scan will be asked to participate.

EXCLUSION CRITERIA

The only exclusion criteria will be subjects with respiratory difficulties.

Children under the age of 12.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Osman MM, Cohade C, Nakamoto Y, Wahl RL. Respiratory motion artifacts on PET emission images obtained using CT attenuation correction on PET-CT. Eur J Nucl Med Mol Imaging. 2003 Apr;30(4):603-6. doi: 10.1007/s00259-002-1024-x. Epub 2003 Jan 21. PMID 12536242